CLINICAL TRIAL: NCT04341519
Title: "Psychological Burden in ICU Survivors of Severe COVID-19 Pneumonia, Their Relatives and Their Healthcare Providers" "Impact Psychologique de l'épidémie COVID-19 Chez Les Patients, Familles et Soignants de Reanimation" "BURDENCOV"
Brief Title: Psychological Burden in ICU Survivors of Severe COVID-19 Pneumonia, Their Relatives and Their Healthcare Providers
Acronym: BURDENCOV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200389
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Corona Virus Infection; Post-traumatic Stress Disorder
MeSH Terms: conditions — Coronavirus Infections; Stress Disorders, Post-Traumatic | interventions — Maslach Burnout Inventory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Family members: * Age>18y
  * Non-opposition to participate to the telephone interviews
  * One family member per patient: the family member the most implicated in the patient's care
    3 groups of Family members will be enrolled in the study corresponding to patients with COVID-19, patients with seasonal flu and patients with community acquired pneumonia (See below). 1 family member per patient will be recruited.
  Interventions: Behavioral: PTSD
- Patients: Patients:
  * Age>18y
  * Admission to the participating ICUs for any cause of acute respiratory failure during the COVID-19 pandemic
  * Having received invasive or noninvasive mechanical ventilation
  * Non-opposition to participate to the telephone interviews.
    3 groups of patients will be enrolled in the study: patients with COVID-19, patients with seasonal flu and patients with community acquired pneumonia.
  * COVID group : Patients admitted to the ICU for acute respiratory failure and having a positive 2019-nCOV RT PCR in a respiratory / nasal swab sample (GROUP COVID-19)
  * Group FLU : patients admitted to the ICU for acute respiratory failure and having a confirmed influenza pneumonia
  * Group CAP (Community-acquired pneumonia) : patients admitted to the ICU for acute respiratory failure and having a clinically or microbiologically documental community acquired pneumonia with negative COVID-19 and Influenza PCRs.
  Interventions: Behavioral: PTSD
- healthcare providers: Two months after the official end of the COVID-19 peak in France, the local investigator will receive a set of 100 questionnaires. He/she will be responsible for proposing survey participation to volunteer healthcare providers. Those who are interested will be given the information letter and the questionnaires in an envelope. Once completed anonymously, they will seal the envelope and give it to the local investigator who will then send us all completed questionnaires by registered post.
  Interventions: Behavioral: Burnout

INTERVENTIONS:
Behavioral: PTSD — family members: post-traumatic stress disorder (PTSD) related symptoms assessed by Impact of Event Scale Revised (IES-R) at 90 days
  Patients:
  post-traumatic stress disorder (PTSD) related symptoms assessed by Impact of Event Scale Revised (IES-R) at 90 days
  Groups: Family members; Patients
Behavioral: Burnout — Symptoms of burnout as assessed by the Maslash Burnout Inventory
  Groups: healthcare providers

SUMMARY:
Coronavirus disease 2019 (COVID-19) is an infectious disease responsible for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). The infection is highly contagious requiring restrictive and stressful measures for patients, family members and ICU healthcare providers. To avoid contagion, patient isolation has become the rule. For patients, these measures add stress to the ICU environment and deprive them of unrestricted family visits. Family members are not only left with fear but also many unanswered questions. In end-of-life situations, many family members are unable to say good-bye and unable to provide support to their loved-one throughout the process. The impact of exclusion or limited inclusion certainly needs to be explored. Moreover, ICU caregivers are having to face new challenges and to work in a unknown situation, juggling with both professional issues such as increased workload, working longer hours and safety issues, and personal issues such as child care and transport as well as family transmission of the virus.

The main objective of this study is to demonstrate that the COVID-19 pandemic, as compared to seasonal flu and community acquired pneumonia, significantly increases post-traumatic stress disorder (PTSD) in family members of critically ill patients.

PTSD-related symptoms will be assessed in family members using the IES-R (impact of event scale revised) during a telephone interview 90 days after ICU discharge. The IES-R is a 22-item self-report measure that assesses subjective distress caused by traumatic events. It will be compared across the three groups (COVID-19, FLU and CAP).

ELIGIBILITY:
Inclusion Criteria:

* Patients:

  * Age>18y
  * Admission to the participating ICUs for any cause of acute respiratory failure during the COVID-19 pandemic
  * Having received invasive or noninvasive mechanical ventilation
  * Non-opposition to participate to the telephone interviews.

Family members:

* Age>18y
* Non-opposition to participate to the telephone interviews
* One family member per patient: the family member the most implicated in the patient's care

Healthcare providers:

* All nurses and physicians (including those in training) in the participating ICUs during the COVID-19 pandemic

Exclusion Criteria:

* Patients:

  * Language barrier to be able to respond to the telephone interview
  * Cognitive disorders disabling patients to respond to the telephone interview
  * Person under legal protection (1121-8 of CSP, Public Health Code) Failure to obtain the non-opposition

Family members:

* Language barrier to be able to respond to the telephone interview
* Person under legal protection (1121-8 of CSP, Public Health Code)
* Failure to obtain the non-opposition

Healthcare providers:

Failure to obtain the non-opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Family members, Patients hospitalized in ICU for COVID19 infection. Healthcare providers involved in care of patients hospitalized in ICU for COVID19 infection.
Sampling Method: Probability Sample
Enrollment: 1464 (Estimated)
Dates: Start 2020-04-06 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
PTSD Family members sup 22 | 90 days
  Proportion of Family members with IES-R> 22 PTSD-related symptoms will be assessed in family members using the IES-R (impact of event scale revised) during a telephone interview 90 days after ICU discharge of corresponding patient. It si a scale ranging from 0 to 88.
  Weiss, DS.; Marmar, CR. The impact of event scale - revised. In: Wilson, JP.; Keane, TM., editors.Assessing psychological trauma and PTSD. New York: Guilford Press; 1997. p. 399-411

SECONDARY OUTCOMES:
PTSD Family members | 90 days
  Among Family members PTSD-related symptoms will be assessed in family members using the IES-R (impact of event scale revised)
PTSD Patients | 90 days
  Among Patients PTSD-related symptoms will be assessed in family members using the IES-R (impact of event scale revised)
PTSD healthcare providers | 2 months after official end of the Covid-19 peak
  Among healthcare providers PTSD-related symptoms will be assessed in family members using the IES-R (impact of event scale revised)
HADS Family members | 90 days
  Among Family members Symptoms of anxiety and depression using the HADS scale
HADS Patients | 90 days
  Among Patients Symptoms of anxiety and depression using the HADS scale
SF36 Patients | 90 days
  Among Patients Mental and physical health-related quality of life as assessed by the SF36
Questionnaire Family members | 90 days
  Among Family members Questionnaire describing their experience of the patient's ICU hospitalization
Questionnaire Patients | 90 days
  Among Patients Questionnaire describing their experience of the patient's ICU hospitalization
Questionnaire healthcare providers | 2 months after official end of the Covid-19 peak
  Among healthcare providers Questionnaire describing their experience of the patient's ICU hospitalization
MBI healthcare providers | 2 months after official end of the Covid-19 peak
  Among healthSymptoms of burnout on MBI scale as assessed by the Maslash Burnout Inventorycare providers
Karasec instrument healthcare providers | 2 months after official end of the Covid-19 peak
  Job Strain as assessed by the Karasec instrument

CONTACTS AND LOCATIONS:
Overall Officials: Elie AZOULAY, MD PhD, Principal Investigator — APHP
Locations (3):
- France (3):
  - Cochin, Paris
  - Pitié Salpetrière, Paris
  - Saint-Louis Hospital, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Azoulay E, Resche-Rigon M, Megarbane B, Reuter D, Labbe V, Cariou A, Geri G, Van der Meersch G, Kouatchet A, Guisset O, Bruneel F, Reignier J, Souppart V, Barbier F, Argaud L, Quenot JP, Papazian L, Guidet B, Thiery G, Klouche K, Lesieur O, Demoule A, Guitton C, Capellier G, Mourvillier B, Biard L, Pochard F, Kentish-Barnes N. Association of COVID-19 Acute Respiratory Distress Syndrome With Symptoms of Posttraumatic Stress Disorder in Family Members After ICU Discharge. JAMA. 2022 Mar 15;327(11):1042-1050. doi: 10.1001/jama.2022.2017. PMID 35179564